CLINICAL TRIAL: NCT05401045
Title: Effect of a Self-designed Metabolic Equivalent Exercise Intervention on Cancer-related Fatigue in Patients With Gastric Cancer
Brief Title: Effect of a Self-designed MET Exercise Intervention on Cancer-related Fatigue in Patients With Gastric Cancer
Acronym: SMEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, lei huang, Research Associate Fellow; PI, Ruijin Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RJHK-2020-16
Record Dates: First submitted 2022-05-15; First posted 2022-06-02 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Neoplasm of Stomach
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observation group (Experimental): 1. Exercise plan: Each session of the self-designed METexercises were divided into 8 components. There are 4 sets and 8-repetitions per component, taking approximately 4 minutes to complete and consuming approximately 18 calories. Patients were instructed to exercise once in the morning and once in the evening.Metabolic equivalent intensity: The intensity of exercise was expressed as metabolic equivalents (METs).
  2. Exercise training: Members of the fatigue management team in the ward taught the patients to perform MET exercises using videos.The fatigue management team members confirmed that the patient could perform the exercise independently and correctly.
  Interventions: Behavioral: Met exercises
- control group (No Intervention): Participants received routine exercise health education that included information pertaining to CRF (causes of CRF, clinical manifestations, related factors, the necessity and importance of fatigue prevention, and measures to improve CRF, etc.) and exercise (3-5 times per week, regardless of the type of exercise). The patients were also informed about the precautions for exercise.

INTERVENTIONS:
Behavioral: Met exercises — Exercise plan: Each session of the self-designed MET exercise program was divided into 8 components: stretching exercises, chest expansion exercises, kicking exercises, lateral movement exercises, body rotation exercises, whole-body exercises, jumping exercises, and a cool down. There are 4 sets and 8-repetitions per component, taking approximately 4 minutes to complete and consuming approximately 18 calories. Patients were instructed to exercise once in the morning and once in the evening. For patients with moderate fatigue and an RPFS score of 4 to 6 points, low-intensity exercise was recommended, i.e., patients could choose 1 to 4 metabolic equivalent exercises and repeat them twice; for patients with mild fatigue and an RPFS score of 1 to 3 points, moderate-intensity exercise was recommended, i.e., patients could choose to complete the entire set of metabolic equivalent exercises or 5 to 8 of the exercises and repeat them twice. The exercise frequency was 5 times per week.
  Arms: observation group

SUMMARY:
To investigate the effect of using Self-arranged Metabolic Equivalent Exercises on cancer-related fatigue in gastric cancer patients. Gastric cancer patients admitted to the oncology department of a tertiary hospital in Shanghai were selected as study subjects and randomly divided into observation group and control group. The experimental group used Metabolic Equivalent Exercises for intervention besides exercise education and implemented records. In the control group, conventional exercise catharsis was performed. The Piper Revised Fatigue Scale (RPFS) and QLQ-30 Quality of Life Scale were used to measure cancer-caused fatigue and quality of life in both groups at the first admission and after 3 months.

DETAILED DESCRIPTION:
This study was a randomized controlled trial. The subjects were randomly assigned into a SMEE or a control group.

For the SMEE group:

1. The general information questionnaire, RPFS, and the Chinese version of the EORTC QLQ-C30 (V3.0) were used for the baseline assessment of patients, and intervention was performed for patients with an RPFS score greater than or equal to 1.
2. Exercise plan: Each session of the SMEE program was divided into 8 components: Stretching exercises, chest expansion exercises, kicking exercises, lateral movement exercises, body rotation exercises, whole-body exercises, jumping exercises, and a cooldown. There were 4 sets and 8 repetitions per component, taking approximately 4 minutes to complete and consuming approximately 18 calories. Patients were instructed to exercise once in the morning and once in the evening. For patients with moderate fatigue and with an RPFS score of 4 to 6 points, low-intensity exercises were recommended, i.e., patients could choose 1 to 4 metabolic equivalent exercises and repeat them twice; for patients with mild fatigue and with an RPFS score of 1 to 3 points, moderate-intensity exercises were recommended, i.e., patients could choose to complete the entire set of metabolic equivalent exercises or 5 to 8 of the exercises and repeat them twice. The exercise frequency was 5 times per week. Nurses informed the participants of the precautions for exercises to ensure safe implementation.

   Metabolic equivalent intensity: The intensity of exercises was expressed as metabolic equivalents (METs). For this study, greater than or equal to 6 METs indicated high intensity, 3 to 5.9 METs moderate intensity, and less than 3 METs low intensity.
3. Exercise training: Members of the Fatigue Management Team in the ward taught the patients to perform metabolic equivalent exercises using videos. Exercise guidance was provided after assessments of surgical, catheter, and incisional pain. Patients could follow the department's WeChat public account to watch complete videos pertaining to metabolic equivalent exercises and related exercise precautions. The Fatigue Management Team members confirmed that a patient could perform the exercise independently and correctly.
4. Health education: The participants were provided with information related to CRF (causes, clinical manifestations, associated factors, the necessity and importance of fatigue prevention, and measures to reduce CRF, etc.) and exercises (intensity, time, frequency, precautions, etc.)
5. Recording: Each participant completed a form after each exercise session.
6. Follow-up: A nurse followed up with each patient by telephone every 2 weeks to determine if the patient completed his or her exercise sessions. Exercise completion rate (%)=(actual exercise time÷planned exercise time)×100%. Nurses supervised and provided reminders to patients with completion rates below 50%. In addition, each patient's exercise success rate was calculated: Exercise success rate (%)=(real-time heart rate after exercise÷target heart rate)×100% (>70% was considered to be up to standard). Target heart rate=(200-age)×100%; a heart rate of 70% to 80% of the target heart rate could improve cardiopulmonary function.

For the control group:

Participants received routine exercise health education that included information pertaining to CRF (causes, clinical manifestations, associated factors, the necessity and importance of fatigue prevention, and measures to reduce CRF, etc.) and exercises (3-5 times per week, regardless of the type of exercises). The patients were also informed of the precautions for exercise.

After 3 months, the SMEE and the control groups were reassessed using the RPFS and the Chinese version of the EORTC QLQ-C30 (V3.0).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Clear pathological diagnosis and staging;
* Undergoing chemotherapy
* CRF based on a total score ≥1 on the revised Piper Fatigue Scale (RPFS) after admission;
* CRF with a Barthel index greater than 80 points;
* Agreed to participate voluntarily and signed an informed consent form;
* Life expectancy of at least 3 months

Exclusion Criteria:

* Patients with heart, lung, liver, kidney and other vital organ failure;
* Patients with mental disorders and unable to communicate verbally;
* Patients with sudden changes in the disease course.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Fatigue state using the Revised Piper Fatigue Scale (RPFS) | up to 3 months
  Cancer-related fatigue is distressing persistent, subjective sense of physical, emotional and/or cognitive tiredness or exhaustion related to cancer or cancer treatment that is not proportional to recent activity and interferes with usual functioning. To use the Revised Piper Fatigue Scale (RPFS) to investigate the fatigue state.The RPFS includes 22 items and 3 open-ended questions regarding the duration of fatigue, the possible causes of fatigue, fatigue-influencing factors, measures to relieve fatigue, and symptoms related to fatigue[7]. The 22 items address the degree that fatigue affects daily activities (6 items), emotional (5 items) and physical (5 items) factors that affect fatigue, and the cognitive and emotional statuses of the respondent (6 items). A number from 0 to 10 is used to indicate the degree of fatigue, with 0 indicating no fatigue and 10 the most severe fatigue; the higher the score is, the more severe the fatigue is.

SECONDARY OUTCOMES:
Quality of life using the European Organization for Research and Treatment of Cancer QLQ-C30 (EORTC-C30) | up to 3 months
  Quality of life refers to a person's feeling of life, is a concept of comprehensive evaluation of the pros and cons of life, usually refers to a result of the development of social policies and plans, mainly refers to the state assessment of individual physical, psychological and social functions. We use the European Organization for Research and Treatment of Cancer QLQ-C30 (EORTC-C30) to measure. The scale has a total of 30 items that are evaluated in 5 functional areas (physical, role, emotional, cognitive, and social dimensions). The higher the functional field and overall scores are, the higher the quality of life of the respondent is; the higher the symptom field scores are, the worse the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Huang, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruifeng Z. The influencing Factors of Cancer-Related Fatigue in gastric cancer patients in perioperative period[D].Dalian：Dalian Medical School,2017
- [Background] Xiaodong X, Xiaoyu Z. Latest progress in cancer-related fatigue: Interpretation of National Comprehensive Cancer Network guidelines for cancer-related fatigue version 1.2018[J]. Chinese Journal of Clinical Oncology, 2018,45(16)
- [Background] Mitchell SA, Beck SL, Hood LE, Moore K, Tanner ER. Putting evidence into practice: evidence-based interventions for fatigue during and following cancer and its treatment. Clin J Oncol Nurs. 2007 Feb;11(1):99-113. doi: 10.1188/07.CJON.99-113. PMID 17441401
- [Background] Lian L, Linhui Z, Mingqin C. Advances in diagnostic and assessment scales for cancer-caused fatigue[J].XinJiang Medicine,2016,46(11):1458-1461,1465
- [Background] So WK, Dodgson J, Tai JW. Fatigue and quality of life among Chinese patients with hematologic malignancy after bone marrow transplantation. Cancer Nurs. 2003 Jun;26(3):211-9; quiz 220-1. doi: 10.1097/00002820-200306000-00006. PMID 12832954
- [Background] Chonghua W, Mingqing C, Canzhen Z et al. The Chinese version of EORTC QLQ-C3 form in evaluation of quality of life for patients with cancer[J].Journal of Practical Oncology,2005,20(4):353-355
- [Background] Hojman P, Gehl J, Christensen JF, Pedersen BK. Molecular Mechanisms Linking Exercise to Cancer Prevention and Treatment. Cell Metab. 2018 Jan 9;27(1):10-21. doi: 10.1016/j.cmet.2017.09.015. Epub 2017 Oct 19. PMID 29056514
- [Background] Kun Y,Min L.Impact of quality nursing service on postoperative rehabilitation of patients with rib fractures combined with pneumothorax[J]. Journal of Clinical Medicine in Practice,2017,21(14):185-186
- [Background] Harvey SB, Overland S, Hatch SL, Wessely S, Mykletun A, Hotopf M. Exercise and the Prevention of Depression: Results of the HUNT Cohort Study. Am J Psychiatry. 2018 Jan 1;175(1):28-36. doi: 10.1176/appi.ajp.2017.16111223. Epub 2017 Oct 3. PMID 28969440
- [Background] Nakano J, Hashizume K, Fukushima T, Ueno K, Matsuura E, Ikio Y, Ishii S, Morishita S, Tanaka K, Kusuba Y. Effects of Aerobic and Resistance Exercises on Physical Symptoms in Cancer Patients: A Meta-analysis. Integr Cancer Ther. 2018 Dec;17(4):1048-1058. doi: 10.1177/1534735418807555. Epub 2018 Oct 23. PMID 30352523
- [Background] Jensen W, Bialy L, Ketels G, Baumann FT, Bokemeyer C, Oechsle K. Physical exercise and therapy in terminally ill cancer patients: a retrospective feasibility analysis. Support Care Cancer. 2014 May;22(5):1261-8. doi: 10.1007/s00520-013-2080-4. Epub 2013 Dec 7. PMID 24317851
- [Background] Blaney J, Lowe-Strong A, Rankin J, Campbell A, Allen J, Gracey J. The cancer rehabilitation journey: barriers to and facilitators of exercise among patients with cancer-related fatigue. Phys Ther. 2010 Aug;90(8):1135-47. doi: 10.2522/ptj.20090278. Epub 2010 Jun 17. PMID 20558566
- [Background] Qiqiong T, Liping G, Ruiping L et al. Physical activity state of cancer - related fatigue patients during malignant tumor chemotherapy period and its influencing factor analysis[J]. Nursing practice and research, 2016,13(13):79-80
- [Background] Pearson EJM, Morris ME, McKinstry CE. Cancer related fatigue: implementing guidelines for optimal management. BMC Health Serv Res. 2017 Jul 18;17(1):496. doi: 10.1186/s12913-017-2415-9. PMID 28720109
- [Background] Ballard-Barbash R, Friedenreich CM, Courneya KS, Siddiqi SM, McTiernan A, Alfano CM. Physical activity, biomarkers, and disease outcomes in cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Jun 6;104(11):815-40. doi: 10.1093/jnci/djs207. Epub 2012 May 8. PMID 22570317
- [Background] Sasso JP, Eves ND, Christensen JF, Koelwyn GJ, Scott J, Jones LW. A framework for prescription in exercise-oncology research. J Cachexia Sarcopenia Muscle. 2015 Jun;6(2):115-24. doi: 10.1002/jcsm.12042. Epub 2015 May 11. PMID 26136187
- [Background] Moore SC, Lee IM, Weiderpass E, Campbell PT, Sampson JN, Kitahara CM, Keadle SK, Arem H, Berrington de Gonzalez A, Hartge P, Adami HO, Blair CK, Borch KB, Boyd E, Check DP, Fournier A, Freedman ND, Gunter M, Johannson M, Khaw KT, Linet MS, Orsini N, Park Y, Riboli E, Robien K, Schairer C, Sesso H, Spriggs M, Van Dusen R, Wolk A, Matthews CE, Patel AV. Association of Leisure-Time Physical Activity With Risk of 26 Types of Cancer in 1.44 Million Adults. JAMA Intern Med. 2016 Jun 1;176(6):816-25. doi: 10.1001/jamainternmed.2016.1548. PMID 27183032
- [Background] Xiao Yue , ZHAO Kun, XUE ming ,et al. Study on the comprehensive goal and index system of Healthy China 2030[J].Health economics research, 2017(4):3-7
- [Result] GLOBOCAN 2020. Estimated number of of new cases of new cases in 2020, China, both sex, alll ages. [EB/OB]https://gco.iarc.fr/today
- [Result] Guilan L, Halin W, Jing Z et al. Cancer related fatigue in nasopharyngeal carcinoma patients during radiation therapy: nursing intervention[J]. Journal of Nursing Science, 2014, 29(8):44-45
- See also: GLOBOCAN 2020 — https://gco.iarc.fr/today